CLINICAL TRIAL: NCT03283995
Title: Hemodynamic Assessment in Cardiogenic Shock Regarding the Etiology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-15; 2017-A00563-50 (Other: n°IDRCB)
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- cardiogenic shock without SCA
  Interventions: Other: Cardiac Volume Monitoring VolumeView; Device: echocardiography
- cardiogenic shock with SCA
  Interventions: Other: Cardiac Volume Monitoring VolumeView; Device: echocardiography
- SCA,
  Interventions: Device: echocardiography
- acute left heart failure with severe alteration of LVEF
  Interventions: Device: echocardiography

INTERVENTIONS:
Other: Cardiac Volume Monitoring VolumeView — hemodynamic measure
  Groups: cardiogenic shock with SCA; cardiogenic shock without SCA
Device: echocardiography — hemodynamic measure

SUMMARY:
The classic physiopathology of cardiogenic shock is explained by a systolic ventricular failure, responsible for a decrease in cardiac output associated with high systemic vascular resistances (SVR). This theory is currently challenged in light of the data collected in the SHOCK study, which assessed outcome of early revascularization versus initial medical stabilization, in cardiogenic shock following myocardial infarction.13 A sub-study highlighted depressed SVR in the population with ischemic cardiogenic shock, related to a systemic inflammatory response syndrome.14 Furthermore, mean FEVG was 30% in the SHOCK trial,13 with a similar distribution with post myocardial infarction heart failure patients without signs of shock.15-19 Thus, alteration of myocardial contractility can be only moderate in cardiogenic shock and isn't the only cause responsible for the hemodynamic instability.20 Recent studies suggest the important roles of the peripheral vascular system and neurohormonal system in the genesis and prolongation of cardiogenic shock.12 Vasodilation caused by nitrous oxide synthase activation27 explains the absence of compensating vasoconstriction observed during the SHOCK trial13, and leads to decreased systemic and coronary perfusion, thus increasing myocardial ischemia and initial ventricular dysfunction. 28,29 Cotter et al. conducted an interesting study of hemodynamic evaluation of various cardiac conditions where they observed a significant variability in the peripheral vascular status, with systemic vascular resistances collapsed in certain patients (similar to those observed in septic shock) and rather close to normal or very high resistances in other patients.21 However these data were obtained from a selected group of patients without differentiating the etiology of cardiogenic shock. Finally, the majority of available studies were limited to cardiogenic shock whose etiology was myocardial infarction.

Therapeutic management of cardiogenic shock is based in first intention on an inotropic support by Dobutamine.11,23 However, better outcomes on contractility and microcirculatory state have been observed with the use of a vasopressor support by Norepinephrine, suggesting the importance of SVR decreasing in genesis of cardiogenic shock.14,24 Recent reviews showed very few data on inotropic treatment and association with vasopressor support,22 hence the low level of recommendations in current guidelines.11,23

So far it is crucial to accurately characterize hemodynamic status and in particular the systemic vascular resistance for patients with cardiogenic shock. Important variabilities in hemodynamic profiles observed in Cooter's trial could explain the difficulty in defining an optimal therapeutic strategy.

the investigators hypothesize that the hemodynamic profile, particularly SVR, of patients with cardiogenic shock is different depending on their etiology. Ischemic cardiogenic shock should be characterized by lower SVR, in relation to a major role of systemic inflammatory response syndrome. On the contrary, non-ischemic cardiogenic shock could be associated with normal or elevated SVR, and thus could explain the variability in distribution of SVR.

ELIGIBILITY:
Inclusion Criteria:

* Persistent hypotension (systolic blood pressure <90 mmHg for at least 30 minutes or need for vasopressor support)
* Signs of visceral hypoperfusion (confusion, marbling, oliguria, hyperlactataemia), 11
* Lower heart rate (<1.8 L / min / m2) Adap Suitable or high filling pressures12

Exclusion Criteria:

* Pregnant or nursing women
* Major under guardianship
* Person staying in a health or social facility
* Non-beneficiaries of a social security scheme
* Persons deprived of liberty
* No one is able to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cardiogenic shock.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Monitoring by transpulmonary thermodilution (VolumeView | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assisatnce Publique Hopitaux de Marseille, Marseille, France